CLINICAL TRIAL: NCT01959776
Title: Asymmetrical Recovery of Cone Outer Segment Tips and Foveal Displacement After Macular Hole Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kyorin University (Other)
Responsible Party: Principal Investigator, Makoto Inoue, Associate professor of Ophthalmology, Kyorin University
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: Kyorineye013; Kyorineye013 (Other: Kyorin Eye Center)
Record Dates: First submitted 2013-10-07; First posted 2013-10-10 (Estimated); Last update posted 2013-10-10 (Estimated); Status verified 2013-10

CONDITIONS: Macular Hole
Keywords: cone outer segment tips line, foveal displacement
MeSH Terms: conditions — Retinal Perforations | interventions — Vitrectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vitrectomy (Other)
  Interventions: Procedure: Vitrectomy

INTERVENTIONS:
Procedure: Vitrectomy

SUMMARY:
Evaluation of asymmetry in recovery of cone outer segment tips and foveal displacement after macular hole surgery

ELIGIBILITY:
Inclusion Criteria:

* The patients with macular hole

Exclusion Criteria:

* The patients with follow-up less than 6 months

Ages: 10 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2009-07; Primary Completion 2009-07 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Optical coherence tomography | one year
  Anatomical evaluation detected with optical coherence tomography after surgical intervention

SECONDARY OUTCOMES:
Visual recovery | one year
  The numbers of the patients with visual recovery after surgical intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Kyorin Eye Center, Mitaka, Tokyo, Japan

REFERENCES:
- [Derived] Itoh Y, Inoue M, Rii T, Ando Y, Hirakata A. Asymmetrical recovery of cone outer segment tips line and foveal displacement after successful macular hole surgery. Invest Ophthalmol Vis Sci. 2014 May 6;55(5):3003-11. doi: 10.1167/iovs.14-13973. PMID 24736052